CLINICAL TRIAL: NCT01973023
Title: Improvement of Chronic Stroke Patients Gait Pattern Following Repetitive Multifocal Botulinum Toxin Injection Sessions in Paretic Lower Limb: an Observational Study.
Brief Title: Stroke's Gait Pattern Modifications of Induced by Repeated BTI
Status: Completed | Type: Observational
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Principal Investigator, Nicolas ROCHE, MDPHD, Centre d'Investigation Clinique et Technologique 805
Other Study IDs: 1687472
Record Dates: First submitted 2013-10-09; First posted 2013-10-31 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2014-03

CONDITIONS: Effect of Repeated Botulinum Toxin Injection on Gait Pattern in Stroke Patients
Keywords: botulinum toxin injection; stroke; 3D motion analysis; gait pattern
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic spastic stroke patients: Chronic spastic stroke patients treated regularly with botulinum toxin injection in lower limb muscles
  Interventions: Other: Motion analysis

INTERVENTIONS:
Other: Motion analysis — Motion analysis was used to assess the modifications of gait pattern in chronic spastic stroke patients regularly treated with botulinum toxin injection

SUMMARY:
Chronic stroke patients exhibit gait pattern alterations which are mainly due to spasticity and treated with repetitive multifocal botulinum toxin injection(BTI). Several studies demonstrated that single BTI-session in a single muscle of paretic lower limb(LL) improved kinematic gait parameters(GP) but surprisingly none of them assessed the effects of repetitive multifocal BTI on patient's gait pattern and their duration.

The aim was to evaluate the impact of repetitive multifocal BTI-sessions on GP of chronic stroke patients. To that end, gait of patients has been compared using 3D-gait analysis after at least 2 consecutive BTI sessions.

DETAILED DESCRIPTION:
All the patients will be tretaed with BTI . these injections will be performed under electrical stimulation control (~5mA). The dose, the number of site of injection per muscle is at the discretion of the physician according to patients' needs and physicians' routine clinical practice. The dilution the most commonly used will depend on the type of BoNT-A (BOTOX®, XEOMIN® or DYSPORT®) and was 100 U for 2.5ml (BOTOX® and XEOMIN®) or 500 U for 2.5 ml (Dysport®).

ELIGIBILITY:
Inclusion Criteria:

->18 years

* a single hemispheric cerebral vascular lesion more than 6 months previously
* able to walk 10 meters without any assistance
* having benefited of at least 2 consecutive BTI sessions, second 3D gait analysis performed at least 3 months after the last BTI.

Exclusion Criteria:

* patient's refusal to participate to the study
* Inability to read the selected text
* Inability to cooperate
* No affiliation to social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: STROKE PATIENTS
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-07; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
kinematics gait parameters | 3h
  peak knee flexion in swing phase(°)

SECONDARY OUTCOMES:
spatiotemporal gait parmeters | 3h
  gait velocity(m/s)

CONTACTS AND LOCATIONS:
Overall Officials: ROCHE Nicolas, MDPHD, Principal Investigator — HOPITAL RAYMOND POINCARE-GARCHES
Locations (1):
- Hopital Raymond Poincare, Garches, Garches, France